CLINICAL TRIAL: NCT02270385
Title: The Effectiveness of a Pressure Ulcer (PU) Prevention Programme for Older People in For-profit Private Nursing Homes (NHs): a Cluster Randomized Controlled Trial
Brief Title: The Effectiveness of a Pressure Ulcer Prevention Programme for Older People in For-profit Private Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Enid Kwong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSEARS20140223001
Record Dates: First submitted 2014-09-16; First posted 2014-10-21 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Prevention of Pressure Ulcers
Keywords: pressure ulcer; nursing home
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group will be implemented a 16-week PU prevention programme. The PU prevention programme includes an intensive training on knowledge and skills ono PU prevention and also a PU prevention protocol. The purpose of the programme is to equip care staff with PU knowledge and skills and to guide especially health workers and personal care workers in PU prevention.
  Interventions: Behavioral: PU prevention programme
- control group (Other): The control group will be provided with the usual PU prevention care
  Interventions: Behavioral: Usual PU prevention care

INTERVENTIONS:
Behavioral: PU prevention programme — The PU prevention programme consists of two major components which are an intensive training course(a 2-hour lecture and two skill training sessions) and a PU prevention protocol.
  Arms: Experimental group
Behavioral: Usual PU prevention care — Usual PU prevention care that is a series of basic nursing care activities: repositioning of residents, moisturization , change of napkins to keep buttock dry.
  Arms: control group

SUMMARY:
This study aims to evaluate the effectiveness of a PU prevention programme for for-profit private nursing homes

DETAILED DESCRIPTION:
The study will be conducted as a two-arm cluster randomized controlled trial, which will compare the efficacy of a PU prevention programme versus usual PU prevention for older people in eight for-profit private nursing homes in Hong Kong. For-profit private NHs recruited will be randomly assigned as experimental or control groups. The nursing homes in the experimental group will be implemented a PU prevention programme. The programme includes a training course which was tailor-made for health workers(HWs) and persona care workers (PCWs) and also a 16-week PU prevention protocol. The outcome measures are incidence and prevalence rate of PUs as well as level of PU knowledge and skill among care staff in the nursing homes. In data analysis, survival analysis will be adopted for identifying PU incidence and prevalence rate. GEE will be used to analyze the time and effect differences of PU knowledge and skills among the care staff between two groups.

ELIGIBILITY:
Inclusion Criteria :

* For-profit private nursing homes having been classified as the category A2 homes in the Enhanced Bought Place Scheme and are eager to improve current pressure ulcer prevention care;
* For for-profit private nursing homes having a capacity of around 130-150 beds;
* For for-profit private nursing homes having no structured PU prevention protocol, and/or programmes in place;- Residents aged 60 or above
* Care staff including personal care workers, health workers and nurses who provide direct care to residents.

Exclusion Criteria:

* Care staffs who are not speak in Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1013 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-09-10 (Actual); Study Completion 2016-09-10 (Actual)

PRIMARY OUTCOMES:
Pressure ulcer incidence | The PUs incidence will be summed up for three periods of time, from T0 to T1, T1 to T2 and T2 to T3.
  The two RAs will inspect the skin of each residents three times a week to detect the first PUs ( those detected on residents without PUs) and the new PUs (those detected on residents already suffering from PUs), starting from one day before the staff training to the end of the protocol implementation (. The numbers, locations, and stages of the PUs detected will be recorded in the PU incidence form. The PU incidence will be then summed up for three periods of time as following. T0 to T1: one day before the commencement of the training course (T0) to the day immediately before the commencement of the protocol implementation (T1) .T1 to T2: the day immediately before the commencement of the protocol implementation (T1) to the eighth week after the commencement of the protocol implementation (T2).T2 to T3: the eighth week after the commencement of the protocol implementation (T2) to the sixteenth week of protocol implementation (T3).

CONTACTS AND LOCATIONS:
Overall Officials: Enid Kwong, PhD, Principal Investigator — Tung Wah College
Locations (1):
- Tung Wah College, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwong EW, Chen LY, Kwan RY, Lee PH. The effectiveness of a pressure injury prevention program for nursing assistants in private for-profit nursing homes: A cluster randomized controlled trial. J Adv Nurs. 2020 Jul;76(7):1780-1793. doi: 10.1111/jan.14391. Epub 2020 May 11. PMID 32285486
- [Derived] Kwong EW, Lee PH, Yeung KM. Study protocol of a cluster randomized controlled trial evaluating the efficacy of a comprehensive pressure ulcer prevention programme for private for-profit nursing homes. BMC Geriatr. 2016 Jan 18;16:20. doi: 10.1186/s12877-016-0189-2. PMID 26782677